CLINICAL TRIAL: NCT07055594
Title: A Phase I/IIa Dose-escalation, Dose-optimization and Dose Expansion Study to Evaluate the Safety and Preliminary Efficacy of Tri-specific Antibody (SOA101) in Subjects With Advanced Solid Tumors.
Brief Title: A Study to Investigate Safety and Preliminary Efficacy of SOA101 in Adult Subjects With Advanced Solid Tumors
Acronym: NbTAST-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shine-On Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOA101-CL-Proto-01
Record Dates: First submitted 2025-06-18; First posted 2025-07-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOA101 (Experimental)
  Interventions: Drug: SOA101

INTERVENTIONS:
Drug: SOA101 — Participants will receive SOA101. The RP2D will be determined based on the results of the Phase I study. During the dose expansion phase, participants will receive SOA101 at the RP2D regimen.

SUMMARY:
The investigational drug, SOA101, is a nanobody-based trispecific antibody T cell engager targeting PD-L1/HLA-G/CD3. This is a Phase I/IIa study including dose-escalation, dose optimization and dose expansion parts to exam safety, tolerability, pharmacokinetics, immunogenecity and efficacy of SOA101 on advanced or metastatic solid tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years old.
2. Subjects with locally advanced, or metastatic solid tumors confirmed histologically or cytologically as one of the following cancer types for whom no suitable alternative standard-of-care therapy exists:

   1. Non-small cell lung cancer (NSCLC);
   2. Ovarian cancer (OC);
   3. Head and neck carcinoma (H&N);
   4. Breast cancer (BC);
   5. Colorectal cancer (CRC).
3. Pathologically confirmed combined positive score (CPS) with ≥ 1% expression of PD-L1.
4. At least one measurable lesion
5. Adequate organ function
6. Female subject must either not be of childbearing potential or a negative pregnancy test
7. Non-vasectomized male subjects must practice highly effective contraception

Exclusion Criteria:

1. Active bacterial, fungal, viral OR atypical infection requiring systemic medication.
2. Received any investigational drug within 4 weeks before screening.
3. Confirmed active HIV (without controlled disease on HAART), HBV, or HCV infection.
4. Symptomatic, unstable central nervous system malignancy OR metastasis
5. Have received organ or tissue transplantation or allogeneic cell therapies.
6. Non-adequate cardiac function
7. Known hypersensitivity to any anti-PD-L1 therapy or anti-CD3 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of SOA101 for Phase I | from start until 3 months after the last dosing
Objective Response Rate (ORR) of SOA101 for Phase IIa | from start until 3 months after the last dosing

SECONDARY OUTCOMES:
Area Under the Curve of SOA101 (AUC) | Up to end of study visit (90 days after the last dose)
  Pharmacokinetics (PK) parameters
Maximum observed plasma concentration of SOA101 (Cmax) | Up to end of study visit (90 days after the last dose)
  Pharmacokinetics (PK) parameters
Half-life of SOA101 (T1/2) | Up to end of study visit (90 days after the last dose)
  Pharmacokinetics (PK) parameters
Overall Response Rate (ORR) | Up to end of study visit (90 days after the last dose)
  Evaluation of anti-tumor activity of SOA101

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin YC, Chen MC, Huang SW, Chen Y, Ho JH, Lin FY, Tan XT, Chiang HC, Huang CC, Tu CY, Cho DY, Chiu SC. Targeting Dual Immune Checkpoints PD-L1 and HLA-G by Trispecific T Cell Engager for Treating Heterogeneous Lung Cancer. Adv Sci (Weinh). 2024 Nov;11(41):e2309697. doi: 10.1002/advs.202309697. Epub 2024 Sep 5. PMID 39234811